CLINICAL TRIAL: NCT05892731
Title: Study of Cognitive Reserve Disorder Affecting Depression in Age- Related Hearing Loss Via Rest State EEG
Brief Title: Study of Cognitive Reserve Disorder Affecting Depression in Aged Related Hearing Loss Via Rest State EEG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-424-01
Record Dates: First submitted 2023-05-25; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-01

CONDITIONS: Age-related Hearing Loss; Cognitive Decline; Depression
MeSH Terms: conditions — Presbycusis; Cognitive Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- age-related hearing loss with depression: According to Hamilton depression scale, age-related hearing loss patients were divided into two groups, namely age-related hearing loss with depression and age-related hearing loss without depression.
  Interventions: Other: with depression
- age-related hearing loss without depression: According to Hamilton depression scale, age-related hearing loss patients were divided into two groups, namely age-related hearing loss with depression and age-related hearing loss without depression.
  Interventions: Other: without depression

INTERVENTIONS:
Other: with depression — age-related hearing loss with depression
  Groups: age-related hearing loss with depression
Other: without depression — age-related hearing loss without depression
  Groups: age-related hearing loss without depression

SUMMARY:
In this study, patients with aged-related hearing loss with depression and without depression were evaluated by audiometry (pure tone audiometry and speech audiometry), cognitive function assessment (MMSE scale for simple mental state test, MoCA Scale for Montreal Cognitive Assessment), and depressive symptoms assessment (GDS-15 and HAMD), resting state EEG. The ananlysis of resting state EEG included power spectral density, traceability analysis, functional connectivity, microstate, clustering coefficient, characteristic path length, characteristic path permeability, and compatibility coefficient. EEG signals were used to explore the activation of brain regions and poor connectivity of brain regions affected by cognitive reserve dissonance on the level of brain imaging. This paper innovatively explores the influence of cognitive reserve dissonance on depressive mood in senile deafness by means of audiological assessment, cognitive function assessment, depression symptom assessment, resting state electroencephalography (EEG) and other technical means. Auditory and cognitive cortical activation, functional connectivity of brain regions, small-world attributes and microstates were analyzed in senile deafness with or without depression at the brain imaging level.

DETAILED DESCRIPTION:
In this study, patients with aged-related hearing loss with depression and without depression were evaluated by audiometry (pure tone audiometry and speech audiometry), cognitive function assessment (MMSE scale for simple mental state test, MoCA Scale for Montreal Cognitive Assessment), and depressive symptoms assessment (GDS-15 and HAMD), resting state EEG. The ananlysis of resting state EEG included power spectral density, traceability analysis, functional connectivity, microstate, clustering coefficient, characteristic path length, characteristic path permeability, and compatibility coefficient. EEG signals were used to explore the activation of brain regions and poor connectivity of brain regions affected by cognitive reserve dissonance on the level of brain imaging. This paper innovatively explores the influence of cognitive reserve dissonance on depressive mood in senile deafness by means of audiological assessment, cognitive function assessment, depression symptom assessment, resting state electroencephalography (EEG) and other technical means. Auditory and cognitive cortical activation, functional connectivity of brain regions, small-world attributes and microstates were analyzed in senile deafness with or without depression at the brain imaging level.

ELIGIBILITY:
Inclusion Criteria:

* age ≥55 years, < 90 years;
* For patients diagnosed with senile deafness, refering to Expert Consensus on Diagnosis and Intervention of Senile Hearing Loss, 2019 edition.
* mild, moderate, moderate and severe sensorineural hearing loss;
* Chinese who can cooperate with all Chinese version evaluation;
* right-handed;
* there was no middle ear disease or inner ear disease;
* there was no bilateral symmetry or sensorineural deafness;
* there was no severe neurological disease, serious systemic disease, family genetic history, or severe mental disease;
* there was no experience of hearing aids fitting.

Exclusion Criteria:

* pure tone audiometry suggests that the average pure tone hearing threshold (500Hz, 1kHz, 2kHz, 4kHz) is > 91dB HL;
* sensorineural hearing loss caused by noise or drugs.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, PASS 15.0 was used to calculate the sample size, and the number of cases was arranged in a 1:1 ratio. The test efficacy was 1-β = 0.9, the test level was α = 0.05, σ=3.0. 17 cases were required in each group. Considering the 20% shedding rate, 22 cases were required in each group. Consequently, 44 cases of age-related hearing loss were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
score of Montreal Cognitive Assessment scale | 1 day of enrollment
  The Montreal Cognitive Assessment Scale(MoCA) is an assessment tool used to rapidly screen for cognitive abnormalities. The test included 11 tests in eight cognitive areas, including attention and concentration, executive function, memory, language, visual structure skills, abstract thinking, calculation, and orientation. Total score of 30 points, and the score of high school/technical secondary school or below needs to be added 1 point. Level: Normal 26-30 , mild cognitive impairment(MCI) 18-25, moderate cognitive impairment 10-17, severe cognitive impairment 0-9.
score of Mini-mental State Examination | 1 day of enrollment
  Mini-mental State Examination (MMSE) is a scale for screening cognitive impairment and is widely used in dementia screening. The scale is divided into seven aspects, including time orientation, place orientation, immediate memory, attention and gauging, delayed memory, language and visual space. There are 30 items in the scale, with a total score of 30. The scale is 27 to 30 points normal, 21 to 26 points mild cognitive impairment, 10 to 20 points moderate cognitive impairment, and 0 to 9 points severe cognitive impairment.

SECONDARY OUTCOMES:
pure tone average | 1 day of enrollment
  With the national standard of hearing soundproof room, using Denmark international hearing AC40 pure tone audiometer, Hugson-westlake (HW) method was used to test the bilateral air conduction of 125Hz to 8000Hz and bone conduction of 500Hz to 4000Hz. And its average pure tone hearing threshold PTA (the average value of gas conductance at 500Hz, 1000Hz, 2000Hz, 4000Hz) was obtained. Level: normal, PTA≤25dB HL; mild HL, PTA=26-40dB HL; moderate HL PTA=41-55dB HL; moderate to severe, PTA= 56-70dB HL; severe, PTA=71-90dB HL; profound, PTA≥91dB HL(WHO1980)
speech acceptance threshold | 1 day of enrollment
  Speech audiometry is a kind of audiometry which uses standardized speech signals as acoustic stimuli to test the speech recognition ability of subjects. The minimum sound intensity required by the tester to achieve 50% accuracy in the speech test is recorded as the threshold of speech acceptance threshold.
Maximum speech recognition score | 1 day of enrollment
  Speech audiometry is a kind of audiometry which uses standardized speech signals as acoustic stimuli to test the speech recognition ability of subjects. In the test, the maximum accuracy at 30-40dB HL above PTA threshold was recorded as the maximum speech recognition score.
score of 15-item Geriatric Depression Scale | 1 day of enrollment
  15-item Geriatric Depression Scale (GDS-15) scores ≥6 were classified as having depressive mood, 0-5 as having no depressive mood, 6-9 as mildly depressed, and 10-12 as severely depressed mood.
score of HAMD scale | 1 day of enrollment
  For the 24th version of HAMD depression Scale, the total score > 35 May indicate severe depression; 21-35, may be mild to moderate depression; 9-20, suspected depression; < 8 indicates normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No